CLINICAL TRIAL: NCT01948947
Title: Improving Functions in MTBI Patients With Headache by rTMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: F1359-P; H130281 SPiRE rTMS MTBI HA (Other: San Diego VA Healthcare System)
Record Dates: First submitted 2013-09-17; First posted 2013-09-24 (Estimated); Results first posted 2018-03-26 (Actual); Last update posted 2018-03-26 (Actual); Status verified 2018-02

CONDITIONS: TBI (Traumatic Brain Injury)
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transcranial Magnetic Stimulation (Experimental): Active-repetitive transcranial magnetic stimulation (rTMS) at the dorsal lateral prefrontal cortex.
  Interventions: Device: Transcranial Magnetic Stimulation
- Sham Transcranial Magnetic Stimulation (Sham Comparator): Sham rTMS will consist of the same parameters as active, however, the subject will be shielded from the magnetic field of the coil.
  Interventions: Device: Sham Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — Active-repetitive transcranial magnetic stimulation (rTMS) at the dorsal lateral prefrontal cortex.
  Arms: Transcranial Magnetic Stimulation
Device: Sham Transcranial Magnetic Stimulation — Sham rTMS will consist of the same parameters as active, however, the subject will be shielded from the magnetic field of the coil.
  Arms: Sham Transcranial Magnetic Stimulation

SUMMARY:
Due to recent wars in Afghanistan and Iraq, the number of Veteran suffering from Mild traumatic brain(MTBI) injury and PTSD increases rapidly. Headache is one of the most debilitating clinical symptoms in Veteran with MTBI and the cause of it is still not entirely clear. Recently, the use of non-invasive brain stimulation such as repetitive transcranial magnetic stimulation(rTMS) has yielded favorable clinical outcome in a few intractable chronic central pain conditions including headaches. This study aims to 1) assess the effect of rTMS in relieving headache and improving neurophysiological functions; and 2)explore the neuronal mechanisms associated with MTBI related headache and the analgesic effect of rTMS with function magnetic resonance imaging (fMRI).

DETAILED DESCRIPTION:
This study will only be conducted at the Veterans Affair hospital in San Diego.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age between 18 to 50
* History of MTBI based on the clinical diagnostic criteria
* History of headache more than 3 months
* No prior experience of TMS treatment
* Pre-treatment headache intensity M-VAS 30(0-100 scale) and average daily headache NPS 3(0-10 scale)
* At least one headache exacerbation per day
* A normal brain MRI in the past 3 months

Exclusion Criteria:

* Pregnancy
* History of pacemaker implant
* Any ferromagnetic(e.g. bullet fragment, shrapnel, device implant) in the brain or body that will prohibit the patients from having a brain MRI
* History of dementia, major psychiatric diseases, or life threatening diseases
* Presence of any other chronic neuropathic pain states
* History of seizure
* Pending litigation
* Lack of ability to understand the experimental protocol and to adequately communicate in English
* History of chronic headache prior to the incidence of MTBI

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2014-05; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Albert Y Leung, MD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vaninetti M, Lim M, Khalaf A, Metzger-Smith V, Flowers M, Kunnel A, Yang E, Song D, Lin L, Tsai A, Lee R, Golshan S, Leung A. fMRI findings in MTBI patients with headaches following rTMS. Sci Rep. 2021 May 5;11(1):9573. doi: 10.1038/s41598-021-89118-2. PMID 33953315

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Transcranial Magnetic Stimulation | Sham Transcranial Magnetic Stimulation
Started | 14 | 15
Completed | 14 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Transcranial Magnetic Stimulation | Sham Transcranial Magnetic Stimulation | Total
Number analyzed (Participants) | 14 | 15 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.13 (9.39) | 34.43 (7.66) | 35.28 (8.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 12 | 11 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 7 | 5 | 12
  More than one race | 4 | 6 | 10
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Composite Score of Debilitating Headache (Intensity x Duration x Frequency)
Description: The primary outcome time-point measurement will be averaged from each day the subject is enrolled in the study for each of the 3 time point periods: pre-treatment baseline, 1-week follow-up and 1-month follow-up. The results depict change in the composite score: intensity (scale of 0-10) x duration (# of hours) x frequency (# headaches per week). The larger composite score for each subject, the worse the debilitating headaches.
Time Frame: Subjects will have a total of 9 visits over the span of 3 months, the baseline, 1-week follow-up and 1-month follow up will qualify as a time point at which the outcome is measured and averaged.
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Transcranial Magnetic Stimulation | Sham Transcranial Magnetic Stimulation
Number analyzed (Participants) | 14 | 15
percent change from baseline
  1-Week Follow-Up | -55.3 (29.0) | -1.7 (41.2)
  1-Month Follow-Up | -58.4 (24.4) | -10 (59.9)
Statistical Analysis 1: Comparison: Transcranial Magnetic Stimulation vs Sham Transcranial Magnetic Stimulation; Change from Baseline to 1-Week Post-Treatment; Test type: Other; p < 0.0001, ANOVA
Statistical Analysis 2: Comparison: Transcranial Magnetic Stimulation vs Sham Transcranial Magnetic Stimulation; Change from Baseline to 1-Month Post-Treatment; Test type: Other; p < 0.001, ANOVA

2. Primary Outcome: Percent Change in Persistent Headache Intensity
Description: The persistent headache measure was assessed through a daily headache log over the course of the subjects participation in the study and averaged for the time point period of baseline, 1-week and 1-month results. The persistent headache is based on a scale of 0-10, the higher the persistent headache intensity averaged score the worse the persistent headache.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Transcranial Magnetic Stimulation | Sham Transcranial Magnetic Stimulation
Number analyzed (Participants) | 14 | 15
percent change from baseline
  1-Week Follow-Up | -25.3 (16.8) | -1.0 (11.7)
  1-Month Follow-Up | -22.6 (17.7) | -2.3 (14.5)
Statistical Analysis 1: Comparison: Transcranial Magnetic Stimulation vs Sham Transcranial Magnetic Stimulation; Test type: Other; p < 0.001, ANOVA — Change from Baseline to 1-Week post-treatment
Statistical Analysis 2: Comparison: Transcranial Magnetic Stimulation vs Sham Transcranial Magnetic Stimulation; Test type: Other; p < 0.01, ANOVA — Change from Baseline to 1-Month post-treatment

3. Primary Outcome: Percent Change in Persistent Headache Prevalence
Description: The persistent headache prevalence measure was assessed through a daily headache log over the course of the subjects participation in the study and collected at baseline, 1-week and 1-month. The persistent headache is defined as having had 3+ continuous headaches over the course of the time point periods and was coded as either yes or no. The results indicate the percent change in the prevalence of persistent headaches for the subjects at the time points. A larger reduction percent indicates a larger decrease in subjects with those persistent headaches.
Time Frame: Subjects will have a total of 9 visits over the span of 3 months, the baseline, 1-week follow-up and 1-month follow up will qualify as a time point at which the outcome is measured.
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Transcranial Magnetic Stimulation | Sham Transcranial Magnetic Stimulation
Number analyzed (Participants) | 14 | 15
percent change from baseline
  1-Week Follow-Up | -50 (51) | -7 (26)
  1-Month Follow-Up | -57 (52) | -20 (41)
Statistical Analysis 1: Comparison: Transcranial Magnetic Stimulation vs Sham Transcranial Magnetic Stimulation; Test type: Other; p = 0.009, ANOVA
Statistical Analysis 2: Comparison: Transcranial Magnetic Stimulation vs Sham Transcranial Magnetic Stimulation; Test type: Other; p < 0.01, ANOVA — Change in Baseline to 1-month post-treatment

4. Secondary Outcome: Percent Change in Depression Score From Baseline to 1-Week Post-treatment
Description: Subjects assessed how their headaches interfered with their mood through the Hamilton Rating Scale for Depression assessment at baseline, 1-week follow-up and 1-month follow-up. The outcome was measured by adding the score of each question on the assessment and then comparing the averaged scores at the different time points. The larger the depression score, the more severe the depression. A larger percent change in depression score indicates a change in the severity of the depression.
Time Frame: Subjects will have a total of 9 visits over the span of 3 months and 3 of those visits will qualify as a time point at which outcome is measured.
Measure: Mean (Standard Deviation); unit: percent change in score from baseline
Arm/Group | Transcranial Magnetic Stimulation | Sham Transcranial Magnetic Stimulation
Number analyzed (Participants) | 14 | 15
percent change in score from baseline | -14.8 (22.1) | -2.7 (40.3)
Statistical Analysis 1: Comparison: Transcranial Magnetic Stimulation vs Sham Transcranial Magnetic Stimulation; Test type: Other; p = 0.033, ANOVA

ADVERSE EVENTS:
Arm/Group | Transcranial Magnetic Stimulation | Sham Transcranial Magnetic Stimulation
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/15
Other Adverse Events (participants affected / at risk) | 0/14 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes